CLINICAL TRIAL: NCT00527202
Title: Randomized Placebo-controlled Study of the Efficacy of Botulinum Toxin Type A (Botox) in Spontaneous Pain and Allodynia Related to Traumatic Nerve Injury or Postherpetic Neuralgia
Brief Title: Efficacy Study of Botox to Treat Neuropathic Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Ambroise Paré Paris (Other)
Responsible Party: Principal Investigator, Nadine ATTAL, MD PhD coordinator, Hospital Ambroise Paré Paris
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTXneurop-1
Record Dates: First submitted 2007-09-07; First posted 2007-09-10 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Postherpetic Neuralgia; Nerve Trauma
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- botulinum toxin A (Experimental): active treatment arm using botulinum toxin A max 200 U injected into the painful area using SC injections 2 cm apart
  Interventions: Drug: botulinum toxin A
- placebo (Placebo Comparator): saline injection with the same dosages injected using the same procedure as botulinum toxin A
  Interventions: Drug: botulinum toxin A

INTERVENTIONS:
Drug: botulinum toxin A — Botulinum toxin A versus saline in parallel groups
  Other Names: saline (placebo)

SUMMARY:
Objectives : to investigate the analgesic effects and safety of intradermal botulinum toxin A injection in the treatment of focal painful neuropathies (eg, postherpetic neuralgia, nerve trauma)

DETAILED DESCRIPTION:
The study will be randomized, performed in parallel group and double blind versus saline and will include 30 patients. Botulinum toxin injection will be injected intradermally in the painful area (one single injection) following a method adapted from that used in hyperhidrosis. The patients will be followed for 6 months after the injection. Primary outcome will be self-reported pain from the patients diaries. Secondary outcomes will be neuropathic symptoms, quality of life, allodynia to brush and pressure, detection and pain thresholds, proportion of responders, pain relief and clinical global impression. Clinical assessment will take place before injection then at 1 month, 3 months and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* daily pain for at least 6 months of at least moderate intensity clearly attributed to the nerve lesion
* limited area of pain
* mechanical allodynia in the painful area

Exclusion Criteria:

* contraindication to BTXA formulation
* coagulation disorders
* another painful condition
* current major depression
* history of drug or alcohol abuse
* compensation claim or litigation
* facial neuropathic pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2004-06 (Actual); Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Self-reported pain (numerical scales) on patients diaries | prospective
  pain intensity on numerical rating scales

SECONDARY OUTCOMES:
mean pain (VAS) at each visit Quality of life Proportion of responders % pain relief Clinical global impression Assessment of blindedness | prospective
  VAS for pain intensity

CONTACTS AND LOCATIONS:
Overall Officials: Didier BOUHASSIRA, MD, PHD, Study Director — INSERM U 792; Danièle RANOUX, MD, Study Chair — hôpital de Limoges (FRANCE)
Locations (1):
- Hôpital Ambroise Paré, AP-HP, Boulogne-Billancourt, France